CLINICAL TRIAL: NCT04594005
Title: An Open-label, Multi-center Phase IB/II Study of Abemaciclib With Paclitaxel for CDK4/6 Pathway Activated Tumors
Brief Title: CDK4/6 Tumor, Abemaciclib, Paclitaxel
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyo Song Kim, Principal Investigator, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-0091
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- abemaciclib+paclitaxel (Experimental)
  Interventions: Drug: abemaciclib+paclitaxel

INTERVENTIONS:
Drug: abemaciclib+paclitaxel — Phase 1b: About 3-6 patients enrollment is expected at dose level 1, -1 and -2. Dose reduction will be preceded with 3 patients/cohort until the first DLT with 4 weeks' observation. The recommend phase 2 dose (RP2D) will be defined.
  level1: abemaciclib 100mg bid, D1-28 / paclitaxel 80mg/m2, IV. D1, 8, 15 Q 4 weeks level-1: abemaciclib 100mg bid, D1-28 / paclitaxel 70mg/m2, IV. D1, 8, 15 Q 4 weeks level-2: abemaciclib 50mg bid, D1-28 / paclitaxel 70mg/m2, IV. D1, 8, 15 Q 4 weeks
  Phase2: At the RP2D dose level in phase I part, we will expand phase 2 study.

SUMMARY:
Cyclin D-dependent kinases (CDKs) are often activated in human cancer owing to various genetic and epigenetic events. This affects regulatory pathways, and it results in uncontrolled proliferation due to loss of checkpoint integrity. Most tumors show increased activity of CDKs, and this permits escape from senescence during the evolution of malignancy.

Among them, cyclin D-CDK4/6-INK4 pathway alterations accelerate G1 progression which provides proliferative and survival advantage to cancer. Therefore, preclinical data demonstrated inhibition of cyclin D-dependent kinase activity have therapeutic benefit. CDK4/6 controls entry into cell cycle progression by regulating Retinoblastoma protein (Rb). The majority of human cancers are known to retain wild-type Rb. In addition, CDK4 amplification and mutations also noted in several tumors. In Rb retained tumors, CDK 4/6 inhibitors reduced Rb phosphorylation and induced G1 arrest. In previous study, CDK4/6 inhibitor showed antitumor activities in Rb-positive breast and colon cancer cell lines. Rapid tumor regression was also noticed in mouse xenograft model. In CDK4 amplified sarcoma cell lines, knockdown of CDK4 inhibited cancer cell proliferation.

Cyclin D1 acts with CDK4 and CDK6 to phosphorylate Rb and promote cell-cycle progression, and CDK4/6 inhibitor might be effective for the patients with CCND1/2/3 amplification/mutation or CDK 4/6 amplification. Therefore, basket trial (NCT03310879) is ongoing for the patients with genomic alterations in CCND1, CDKN2A, or CDK4. Amplification/mutation of CCND1/2/3 and CDK4/6 occurs in approximately 15-30% of various solid tumors; sarcoma, GBM, melanoma, gem cell tumor, and gynecologic tumors Regarding the more potent synergistic effect, paclitaxel demonstrated a rationale for promising combination partner with CDK 4/6 inhibitors. In non-small cell lung cancer cell lines, synergistic anti-tumor activities were reported with paclitaxel combination. Corollary, we planned to conduct the phase Ib/II trial of abemaciclib and paclitaxel combination in CDK4/6 pathway activated tumors as one subgroup of multi-arms in ongoing basket trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic solid tumors, for which standard therapy proven to provide clinical benefit no longer

  * CDK4/6 activated tumors on next-generation sequencing or FISH (fluorescence in situ hybridization) analyses

    - CCND1, 2, or 3 high-level amplification, CCND1 mutation, or a CCND1 splice variant expected to lead to nuclear retention of cyclin D1 protein

    - CDK4 or CDK6 high-level amplification
    * ECOG performance status of 0 to 1

      * ≥ 19 years of age

        * Subjects with measurable or evaluable disease ⑥ Subjects who meet the following criteria: - Absolute neutrophil count (ANC) ≥ 1500 /µL (*ANC = Neutrophil segs ＋ Neutrophil bands) - Platelet count ≥ 75,000/ µL - Serum creatinine < 1.5 x upper limit of normal (ULN)

          * AST (SGOT) and ALT (SGPT) < 3 x upper limit of normal (ULN) (If there is Liver Metastasis < 5 x upper limit of normal (ULN))
          * Total bilirubin < 1.5 x upper limit of normal (ULN)

            * Provision of written informed consent prior to any study procedure

Exclusion Criteria:

* Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy.

  * Any previous chemotherapy or immunotherapy within 2 weeks or at least 3-5 half-lives for previous chemo/immunotherapy whichever is longer.

    * Any major operation or irradiation within 2 weeks of baseline disease assessment

      * Any clinically significant gastrointestinal abnormalities which may impair intake or absorption of the study drug

        * Previously abemaciclib-exposed patients

          ⑥ Subjects with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms

          ⑦ Other co-existing malignancies or malignancies diagnosed within the last 3 years with the exception of basal cell carcinoma, thyroid cancer or cervical cancer in situ.

          ⑧ Subjects with an uncontrolled major cardiovascular disease (including AMI within 12 months, unstable angina within 6 months, over NYHA class III congestive heart failure, congenital long QT syndrome, 2° or more AV Block and uncontrolled hypertension)

          ⑨ Active infection including hepatitis B, hepatitis C

          ⑩ Pregnant or lactating female

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
overall response rate | 8 weeks
recommend phase 2 dose | during 28 days after 1st dose
  to find the recommend phase 2 dose

SECONDARY OUTCOMES:
adverse event | 1 week
disease control rate | 8 weeks
progression free survival | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea